CLINICAL TRIAL: NCT00473603
Title: Effect of Free Fatty Acids on Androgen Precursors in Vivo in Healthy Young Women
Brief Title: Effect of Free Fatty Acids (FFA) on Androgen Precursors in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Professor Joachim Spranger, professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201-05
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Hyperandrogenism; Glucocorticoid Metabolism
Keywords: androgens; fatty acids
MeSH Terms: conditions — Hyperandrogenism | interventions — Lipids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LHI (Experimental): to perform an i.v. lipid heparin infusion for 4 h
  Interventions: Drug: lipid/heparin infusion
- SHI (Sham Comparator): to perform an i.v. saline heparin infusion for 4 h
  Interventions: Drug: lipid/heparin infusion

INTERVENTIONS:
Drug: lipid/heparin infusion — to perform an i.v. lipid heparin infusion infusion for 4 h

SUMMARY:
The purpose of this study is to determine whether free fatty acids modify the androgen levels in healthy young women.

DETAILED DESCRIPTION:
Free fatty acids (FFA) are known to play an important role by inducing insulin resistance and metabolic disturbances in obesity and type 2 diabetes. In addition, FFAs seems to have a stimulatory effect on adrenal androgen precursors in men. However, the effect of FFAs on androgen precursors and androgens in women is yet unknown.

Therefore the effect of increased FFAs on adrenal androgens and androgen precursors should be investigated in a randomized controlled cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women

Exclusion Criteria:

* diabetes mellitus or impaired glucose tolerance
* clinical signs of hyperandrogenism
* polycystic ovary
* hormonal therapy
* BMI > 30 kg/m2
* dysmenorrhoea

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
change of DHEA | 1 day
  Measurement of serum DHEA
change of DHEAS | 1 day
  Measurement of serum DHEAS
change of testosterone | 1 day
  Measurement of serum testosterone
change of androstenedione | 1 day
  Measurement of serum androstenedione

SECONDARY OUTCOMES:
urinary androgen excretion | 1 day
urinary cortisol excretion | 1 day
  measurement of urinary cortisol, aTHF and THF
urinary cortisone excretion | 1 day
  measurement of urinary cortisone and THE
changes in metabolic parameters (e.g. FGF-21) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mai, MD, Principal Investigator
Locations (1):
- Charite, Campus Benjamin Franklin, Berlin, Germany